CLINICAL TRIAL: NCT04627272
Title: An Evaluation of the Accuracy of AutoDx-DR, a Software Algorithm That Detects Diabetic Retinopathy From Retinal Images of Individuals With Diabetes
Brief Title: AutoDx-DR Prospective Clinical Validation Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hill-Rom (Industry)
Collaborators: Rho, Inc. (Industry); ClinEdge (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 60095127
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: This is a study to determine the accuracy of AutoDX. All eligible study participants will have a retinal fundus image taken which is then uploaded to the RetinaVue Network. Subjects will also undergo further retinal fundus imaging: four mydriatic, stereoscopic 45° field of view (4W) retinal images and spectral domain optical coherence tomography (SD-OCT) captured with the Reference Standard Camera.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- AutoDX and Gold Standard (Experimental): A licensed clinician will obtain 60° wide single-field retinal fundus images from subjects who are diabetic patients in primary care environments (i.e. non-eye care settings, such as internal medicine, family medicine, and endocrinology). The fundus images will be uploaded to the RetinaVue Network software using the AutoDx-DR with Over-read modality, where images are transmitted to both AutoDx-DR and a remote ophthalmologist. Subjects participating in this study will undergo further retinal fundus imaging: four mydriatic, stereoscopic 45° field of view (4W) retinal images and spectral domain optical coherence tomography (SD-OCT) captured with the Reference Standard Camera
  Interventions: Device: AutoDX-DR

INTERVENTIONS:
Device: AutoDX-DR — AutoDx-DR provides basic image interpretation for the detection of DR and diabetic macular edema (DME) and a Refer or Not Refer recommendation.

SUMMARY:
In this study, we will prospectively evaluate the accuracy of a deep-learning based software algorithm in the detection of diabetic retinopathy from 60° wide single-field retinal fundus images.

DETAILED DESCRIPTION:
We will obtain 60° wide single-field retinal fundus images from subjects who are diabetic patients in primary care environments (i.e. non-eye care settings, such as internal medicine, family medicine, and endocrinology). The fundus images will be uploaded to the RetinaVue Network software using the AutoDx-DR with Over-read modality, where images are transmitted to both AutoDx-DR and a remote ophthalmologist. AutoDx-DR will generate an initial Refer or Not Refer recommendation and the remote ophthalmologist will provide a detailed diagnostic image interpretation which will be used for patient management and referral during the course of the study. AutoDx-DR can also generate a third output which is "Inadequate for Interpretation". In this case, the images will still be sent to the remote ophthalmologist for interpretation. If the ophthalmologist also cannot interpret the images, the patient will be recommended to have an in-person comprehensive ophthalmologic exam.

Subjects participating in this study will undergo further retinal fundus imaging: four mydriatic, stereoscopic 45° field of view (4W) retinal images and spectral domain optical coherence tomography (SD-OCT) captured with the Reference Standard Camera (i.e. Zeiss Cirrus 600 photo, or other appropriate FDA-cleared imaging device with stereo fundus photography and SD-OCT capability that meets the requirements of the certified fundus photography reading center such as Topcon, Optovue, and Heidelberg). The 4W and SD-OCT imaging will be performed by a certified technician located at or near the enrolling study site. The 4W and SD-OCT images will be interpreted by a certified fundus photography reading center (FPRC) for more than mild DR or any diabetic macular edema. The FPRC's Not Refer/Refer determination will be used as the "gold standard" interpretation in this study.

The AutoDx-DR interpretation of the 60° wide single-field images will be compared to the FPRC "gold standard" interpretation for the Not Refer/Refer recommendation. Accuracy metrics of sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR), and negative likelihood ratio (NLR), with 95% confidence intervals will be calculated. All diabetic patients who are attending routine primary care or endocrinology appointments and meet the enrollment criteria will be invited to participate in the study. All study procedures will be performed during a single study visit.

ELIGIBILITY:
Inclusion Criteria:

A documented diagnosis of diabetes mellitus in accordance with the criteria established by the American Diabetes Association (ADA)7 as indicated by at least one of the following:

* Hemoglobin A1c (HbA1c) > 6.5%
* Fasting Plasma Glucose (FPG; period of fasting must be at least 8 hours) > 126 mg/dL (7.0 mmol/L)
* Oral Glucose Tolerance Test (OGTT) with 2-hour plasma glucose >200 mg/dL (11.1 mmol/L), using the equivalent of an oral 75 g anhydrous glucose dose dissolved in water o Symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dL (11.1 mmol/L)

  * 22 years of age or older
  * Ability to understand the study and sign the informed consent

Exclusion Criteria:

* A documented diagnosis of more than mild diabetic retinopathy in the patient record.

  o More than mild diabetic retinopathy shall be defined as moderate NPDR, severe NPDR, proliferative diabetic retinopathy (PDR) or any level of DME; or a documented diabetic eye exam report indicating more than microaneurysms [i.e. presence of intraretinal hemorrhages, venous beading, intraretinal microvascular abnormalities (IRMA,) neovascularization or DME.]
* They report having severe vision loss in both eyes.
* They report a history of laser treatment or surgery of the retina.
* They report that they are currently receiving treatment for DR or DME.
* They report a diagnosis of angle closure glaucoma.
* They report hypersensitivity to light which makes retinal imaging uncomfortable.
* They are currently pregnant or breastfeeding.
* They report that they have an iris supported intraocular lens or anterior chamber intraocular lens associated with a previous cataract surgery.
* They had a previous pupilloplasty surgery.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1539 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Each subject will only have one day study visit and will provide the AutoDX-DR and gold standard reading during their one visit.
  The ability of AutoDX-DR to correctly identify those with the disease (true positive rate)
Specificity | Each subject will only have one day study visit and will provide the AutoDX-DR and gold standard reading during their one visit.
  The ability of AutoDX-DR to correctly identify those without the disease (true negative rate)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Piñero-Piloña, MD, Principal Investigator — Diabetes Care Center; Joseph Woolley, MD, Principal Investigator — Southwest Internal Medicine; Keila Hoover, MD, Principal Investigator — Hoover Family Medicine; Quang Vo, MD, Principal Investigator — Dr. Steven Barag, DO; Peter Mattar, MD, Principal Investigator — Dr. Peter N. Mattar, MD; Efrain Soto, MD, Principal Investigator — Park Lakes Family Medicine; Harish Thakkar, MD, Principal Investigator — Southwest Medical Clinic; Luis Gonzalez-Orozco, MD, Principal Investigator — Clinic of Luis Gonzalez; Jennifer Bellucci-Jackson, MD, Principal Investigator — Family Medicine Specialists

IPD SHARING:
Plan to Share IPD: No